CLINICAL TRIAL: NCT05817487
Title: Effects of Crossover Point Exercise and High-intensity Interval Training on Vascular Health in Young Overweight Females
Brief Title: Effects of COP Exercise and HIIT on Vascular Health in Young Overweight Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EOCPEAHITOVHIYOF
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Experimental)
  Interventions: Behavioral: high-intensity interval training (HIIT)
- COP group (Experimental)
  Interventions: Behavioral: crossover point(COP) exercise training

INTERVENTIONS:
Behavioral: high-intensity interval training (HIIT) — Participants in both the COP and HIIT groups underwent 30 sessions of exercise performed over 10 weeks. The training sessions in the HIIT group involved five high-intensity intervals of 4 minutes each (running or walking on a treadmill) at 85% VO2max interspersed with 3 minutes of low-intensity walking.
  Arms: HIIT group
Behavioral: crossover point(COP) exercise training — Participants in both the COP and HIIT groups underwent 30 sessions of exercise performed over 10 weeks. The COP exercise training sessions involved 45 minutes of continuous exercise at the COP on a treadmill.
  Arms: COP group

SUMMARY:
The goal of this study is to determine the effects of high-intensity interval training and crossover point exercise training on vascular health in young overweight women.

DETAILED DESCRIPTION:
In recent years, improving cardiovascular health through exercise has become a popular research question, however, it is not clear which intensity and modes of exercise bring more benefits. Crossover point(COP) intensity has great medical potential as a personalized exercise intensity that is based on substrate utilization mode, especially in overweight and obese people.On the other hand, several studies have demonstrated that HIIT is an effective method in improving vascular endothelial dysfunction. During our study, we evaluated the vascular health changes in young overweight women who received either COP exercise or HIIT exercise for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-30 years old
2. Body mass index (BMI) < 28 kg/m2 and ≥ 24 kg/m2
3. No exercise habit, and no recent new exercise plan
4. No contraindications to exercise

Exclusion Criteria:

1. Participates had an orthopedic or other condition that limited participation in daily exercise
2. Participates had a history of myocardial infarction, stroke, diabetes mellitus, chronic respiratory disease or cancer
3. Participates had smoking or alcohol behavior

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
brachial-ankle pulse wave velocity (baPWV) | 10 weeks
  The change of baPWV before and after intervention
blood pressure | 10 weeks
  The change of blood pressure before and after intervention

SECONDARY OUTCOMES:
Interleukin 6 (IL-6) | 10 weeks
  The change of IL-6 level before and after intervention
Homocysteine (HCY) | 10 weeks
  The change of HCY level before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, China